CLINICAL TRIAL: NCT03039647
Title: Insulin Resistance and Accelerated Cognitive Aging
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natalie Rasgon, Professor of Psychiatry and Behavioral Sciences, Stanford University
Other Study IDs: 38733
Record Dates: First submitted 2017-01-26; First posted 2017-02-01 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Entry Point IR (SSPG, HOMA-IR): All subjects will undergo baseline indirect (HOMA-IR) and direct (SSPG) measures of IR. The investigators hypothesize that a higher entry point IR will predict steeper decline in memory and executive function performance and hippocampal connectivity.
- Change in IR (HOMA-IR): The investigators predict that change in IR (as measured by HOMA-IR) will predict the pattern of decline in memory and executive function performance and hippocampal connectivity.

SUMMARY:
Premature and accelerated brain aging trajectories have been observed among people with metabolic dysfunction, but mechanisms of these altered trajectories are not understood. Insulin resistance (IR) is known to change with age and affect cognition in older and elderly adults as well as in patients with mood disorders. The main purpose of the study is to describe the developmental trajectory of cognitive and neural biomarkers across the spectrum of metabolic dysfunction in overweight/obese adults younger than 50 years of age. The innovative study design will allow the investigators to examine cognitive outcome development over a 25-year span without an investment into the longitudinal observation of changes in cognition and neural function.

DETAILED DESCRIPTION:
Premature and accelerated brain aging trajectories started to be recognized in cognitive and neural responses, but specific mechanisms for the course of cognitive aging remain to be elucidated. Insulin resistance (IR) is known to change with age, affect cognition in older and elderly adults as well as in patients with affective disorders. It is unknown whether IR can predict cognitive decline in individuals younger than age 50 without overt mental illness. Studies in younger adults afford a unique opportunity to assess whether IR mediates cognitive and correlating neural processes decades before the manifestation of cognitive decline. The investigators propose to use an innovative accelerated longitudinal design (ALD) to characterize trajectories of cognitive and neural biomarkers and to: 1) describe baseline cognitive and neural biomarkers of brain function across the spectrum of IR in persons ages 25-50; 2) assess how the baseline IR and change in IR at a younger age affects the pattern of decline in cognitive and neural biomarkers and 3) explore the effects of baseline IR on changes in cognitive and neural variables of interest as moderated by non-modifiable risk factors for cognitive decline (gender, and APOE4/family history of AD). The current proposal aims to describe the developmental trajectory of cognitive and neural biomarkers across the spectrum of metabolic dysfunction in overweight/obese adults younger than 50 years of age. Utilizing an accelerated longitudinal design (ALD) we will recruit overweight/obese individuals (total N=160) aged 25-50. Based on semi-longitudinal data, this design will allow us to examine outcome development over 25 years between ages 25-50 after 3-year follow-up. All subjects will undergo baseline qualitative measure of IR, cognitive assessments and multimodal magnetic resonance imaging (MMRI). Neuropsychological evaluation will focus on cognitive flexibility/set shifting tests reflecting hippocampal connectivity to the medial prefrontal region. MMRI will include memory-related hippocampal function and connectivity (measured with task- and resting-state fMRI) and hippocampal volumes. The ALD design will allow investigation of the relation between cognitive performance and a corresponding neural response across the IR spectrum over a long period of time and the predictive value of IR of long-term trajectories of change in cognitive and neural biomarkers over span of 25 years.

ELIGIBILITY:
Inclusion Criteria:

* Between 25 and 50 years of age
* BMI of 25 to 33 kg/m^2
* At least 12 years of education
* All subjects will be medically stable (i.e. no uncontrolled or poorly controlled medical illnesses), cognitively intact as defined by Mini Mental Status Exam (MMSE) score of > 27, and will have adequate visual and auditory acuity to allow for cognitive testing. Glycemic history will be collected together with other pertinent medical information from primary care providers.

Exclusion Criteria:

* Diagnosis of possible or probably dementia, MCI, or any other dementia
* Evidence of cognitive decline by MMSE < 27 or self-reported significant decline in memory within the past year (per the Memory Function Questionnaire)
* History of Type 1 or Type 2 Diabetes
* Fasting plasma glucose > 126 mg/dL
* History of significant cardiovascular disease or myocardial infarction, cerebrovascular/pulmonary disease, cancer, untreated hypothyroidism, unstable or untreated hypertension, history of head trauma, MRI-contraindications (i.e. metal in body, claustrophobia), premature birth (which may affect MRI findings), history of neurological disorder (ischemic attacks, carotid bruits, or lacunes upon MRI scan), or evidence of neurological or other physical illness that could produce cognitive deterioration
* Use of any drug that may significantly affect the SSPG or cognitive testing results (specifically: centrally active beta-blockers, narcotics, clonidine, antipsychotics, benzodiazepines, systemic corticosteroids, medications with significant cholinergic or anticholinergic effects, anti-convulsants, anti-diabetics, or anti-cholesterol medications)
* Drug or alcohol abuse or dependence within the past 6 months, or positive urine toxicology screen for illicit substances at eligibility screening
* History of mental illness, with the exception of past mood disorder, or evidence of acute depression as determined by a 17-item Hamilton Depression Rating Scale (HDRS-17) score of 8 or more
* Participants with history of mood disorder must be in remission for at least 6 months prior to study entry

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The investigators will consent and enroll 160 medically stable men and women in and around Stanford. Stanford will be the only study site. Subjects will be 25-50 years old, with a body mass index (BMI) of 25 to 35kg/m2, and will have at least 12 years of education.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in hippocampal connectivity | Change in hippocampal connectivity from entry point to exit point three years later
  This will be assessed by MRI and cognitive assessments.

SECONDARY OUTCOMES:
Change in hippocampal volume | Change in hippocampal volume from entry point to exit point three years later
  This will be determined by MRI analysis.
Change in memory-related functional activation | Change in memory-related functional activation from entry point to exit point three years later
  This will be determined by MRI analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Rasgon, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Psychiatry Building, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No